CLINICAL TRIAL: NCT05725785
Title: Technology-Assisted Implementation of a Mobile Health Program for Serious Mental Illness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Dror Ben-Zeev, Professor, School of Medicine: Psychiatry, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00016266; DI-2021C3-24542 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2023-01-26; First posted 2023-02-13 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-08

CONDITIONS: Schizophrenia; Bipolar Disorder; Major Depressive Disorder; Schizo Affective Disorder
Keywords: serious mental illness; mHealth; digital health; schizophrenia; implementation; smartphone; SMI
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Depressive Disorder, Major; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FOCUS participants (Other): FOCUS is a smartphone application system designed to improve illness self-management and facilitate recovery in individuals with serious mental illness. It delivers both system initiated (i.e. pre-programmed) and patient initiated (i.e. on demand) real-time assessment to individuals in their own environment.
  Interventions: Behavioral: FOCUS participants

INTERVENTIONS:
Behavioral: FOCUS participants — Participants using FOCUS will be given access to the FOCUS application and trained by the mHealth support specialist on how to use the functions of the smartphone (i.e. using a touchscreen, call, text) and different features of the FOCUS intervention.

SUMMARY:
The goal of this clinical trial is to learn about how a digital training platform can enhance implementation and effectiveness of a validated mHealth system, called FOCUS, in people with serious mental illness. The main question this research aims to answer is whether patients obtain similar outcomes to previous FOCUS studies when using FOCUS with clinicians trained on a newly developed digital training platform.

Participants will be asked to use the FOCUS smartphone application and receive mobile health coaching from clinicians who have been trained using the digital training platform.

DETAILED DESCRIPTION:
Widely available technologies can help overcome the capacity constraints of brick-and mortar community mental health centers (CMHCs), expand the reach of evidence-based mental healthcare, and provide much needed illness management skills and resources for people with serious mental illness (SMI). With funding from the NIMH, PCORI, and CMMI, the investigators developed and tested FOCUS--a multi-modal smartphone illness self-management system that is shown to be feasible, usable, highly engaging, and effective among people with SMI.

The current project facilitates translation of FOCUS into routine care at CMHCs using implementation strategies of practice facilitation, implementation resource teams, and the development of accessible training materials. The investigators are proposing a technology-assisted training and implementation model designed to address system needs that have emerged since the COVID-19 pandemic and enhance sustainability of FOCUS at CMHCs. The new tools and strategies used in the project will facilitate improved training and implementation in new treatment settings, reaching a far larger number of patients who otherwise would not receive FOCUS and improving the sustainability of this tool, even in high turnover settings.

This trial is a prospective multi-site site single arm implementation study in three community mental health centers located in New Hampshire and Missouri. The investigators will develop and evaluate a digital training platform to aid in the implementation of FOCUS and utilize the platform to improve the availability, reach, impact, and sustainability of the FOCUS intervention in CMHCs. Patient participants will utilize FOCUS for a 12-week period at CMHCs where clinicians have been trained using the digital training platform. Investigators will compare patient outcomes to results of previous trials where clinicians were trained using more traditional, in-person training and support methods.

ELIGIBILITY:
Inclusion Criteria:

* Chart diagnosis of a serious mental illness (i.e., schizophrenia, schizoaffective disorder, bipolar disorder, major depressive disorder)
* 18 years of age or older
* English-speaking
* Have access to a smartphone that can support FOCUS

Exclusion Criteria:

• Plan to move or discontinue services at the participating community mental health center in the next three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in psychiatric functioning | Baseline, 3-months
  Change in the psychiatric functioning will be measured by the Symptom Checklist-9 (SCL-9). This nine-item questionnaire is used to assess psychiatric functioning with a maximum score of 36 and a minimum score of 0. Higher scores on this scale indicates worse functioning.
Change in depressive symptoms | Baseline, 3-months
  Change in the depressive symptoms will be measured by the Beck Depression Inventory-2 (BDI-2). This 21-item questionnaire is used to assess depressive symptoms with a maximum score of 63 and a minimum score of 0. Higher scores on this scale indicates worse functioning.
Change in auditory verbal hallucinations | Baseline, 3-months
  Change in the auditory verbal hallucinations will be measured by the Hamilton Program for Schizophrenia Voices (HPSVQ). This 13-item questionnaire is used to assess auditory verbal hallucinations with a maximum score of 36 and a minimum score of 0. Higher scores on this scale indicate worse functioning.
Change in recovery oriented thinking | Baseline, 3-months
  Recovery of patient will be measured using the Recovery Assessment Scale (RAS). RAS has 24-items that assess 5 factors related to recovery including Hope, Goal Directedness, and Domination by Symptoms. The maximum score on this scale is 120 and the minimum score is 24. A higher score on this scale indicated improved functioning.
Change in perceived quality of life | Baseline, 3-months
  Quality of Life will be assessed using a 6-item Quality of Life scale of general wellbeing, interpersonal relations, participation in activities, and role functioning. Patients respond on a 7-point scale with a maximum score of 42 and a minimum score of 6. A higher score on this scale indicated a higher quality of life.
Patient Satisfaction with FOCUS | 3-months
  Patient satisfaction related to their use of the FOCUS system will will be assessed by a 5-item questionnaire on a 7-point scale asking about..... The maximum score on this scale is and the minimum is 35 and the minimum score on this scale is 5. A higher score on this scale indicates higher satisfaction with the FOCUS system.
Patient Engagement with FOCUS | 3-months
  Patient engagement will be the number of weeks FOCUS was used, during the 12-week intervention period. Data for FOCUS usage will be captured automatically on FOCUS software.

CONTACTS AND LOCATIONS:
Overall Officials: Dror Ben Zeev, PhD, Principal Investigator — University of Washington
Locations (3):
- United States (3):
  - Places for People, St Louis, Missouri
  - Community Partners, Dover, New Hampshire
  - The Mental Health Center of Greater Manchester, Manchester, New Hampshire

IPD SHARING:
Plan to Share IPD: No